CLINICAL TRIAL: NCT06206642
Title: Evaluation of a Novel Targeted Molecular Probe 18F-FAPI-04 PET/CT for Various Malignant Tumors: Comparison With 18F-FDG PET/CT
Brief Title: Comparing 18F-FAPI-04 and 18F-FDG PET/CT in Cancer Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Xiaoxue Tian, Attending physician, Lanzhou University Second Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: XTian
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Malignant Neoplasm
Keywords: 18F-FDG; 18F-FAPI; PET/CT
MeSH Terms: conditions — Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 18F-FAPI-04 (Experimental): 18F-FAPI-04 PET-CT is injected through the patient's elbow vein without special preparation at a dose of 2.96-5.55 megabecquerels (MBq) /kg (0.08-0.15 millicurie/kg).
  Interventions: Diagnostic Test: PET/CT
- 18F-FDG (Experimental): Before the 18F-FDG PET/CT examination, all patients should fast for at least 4-6 hours, and the fasting blood glucose should be controlled to less than 9.0mmol/L to avoid difficulties in image analysis due to poor blood glucose in patients. 18F-FDG is administered via the patient's elbow vein at a dose of 2.96-5.55 megabecquerels (MBq) /kg (0.08-0.15 millicurie/kg).
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — Low-dose CT images were first collected during scanning. The tube voltage was 120kilovolt, the tube current was 50-220Milliampere and the layer thickness was 3.75mm.

SUMMARY:
Evaluating fluoro-18-fibroblast activation protein inhibitor-04 positron emission computed tomography's diagnostic efficacy for primary malignancies versus 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose.

DETAILED DESCRIPTION:
In recent years, radionuclide labeled fibroblast activating protein inhibitors (FAPIs) have gradually become a new strategy for targeted diagnosis and therapy. In this study, radionuclide 18F was used to label FAPI, and the imaging value of FAPI was compared with that of common developer 18F-FDG. To evaluate the diagnostic value of 18F-FAPI-04 PET/CT in various malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥18 years old); PET/CT examination is required after evaluation by oncologist. Healthy persons who volunteer for PET/CT scans; Can cooperate to complete the inspection process; I or family members, legal representatives agree to participate in the study and can sign the informed consent in person.

Exclusion Criteria:

The patient has a serious underlying disease or mental illness and is unable to cooperate with the PET/CT examination; Have received systematic chemotherapy; Previous history of primary tumor; Pregnancy; I or family members, legal representatives are unable or unwilling to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, accuracy, positive predictive value and negative predictive value of 18F-FAPI-04 PET/CT | 1 week
  McNemar test

CONTACTS AND LOCATIONS:
Overall Officials: Liu Jiangyan, Study Director — Lanzhou University Second Hospital
Locations (1):
- The Second Hospital of Lanzhou University, Lanzhou, Gansu, China